CLINICAL TRIAL: NCT00681941
Title: An Open Label, Dose Titration of Sevelamer Carbonate Tablets Dosed Three Times a Day in Hyperphosphatemic Chronic Kidney Disease Patients Not On Dialysis
Brief Title: An Open Label Dose Titration of Sevelamer Carbonate Tabs 3 Times a Day in Hyperphosphatemic CKD Patients Not On Dialysis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Genzyme, a Sanofi Company (Industry)
Responsible Party: Medical Monitor, Genzyme Corporation
Organization: Sanofi (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SVCARB00105; ACTRN012606000380594
Record Dates: First submitted 2008-05-19; First posted 2008-05-21 (Estimated); Last update posted 2015-03-20 (Estimated); Status verified 2015-03

CONDITIONS: Chronic Kidney Disease; Hyperphosphatemia
MeSH Terms: conditions — Renal Insufficiency, Chronic; Hyperphosphatemia | interventions — Sevelamer

ARMS (1):
- 1 (Experimental): Sevelamer Carbonate Tablets Dosed Three Times A Day
  Interventions: Drug: Sevelamer carbonate (Renvela®)

INTERVENTIONS:
Drug: Sevelamer carbonate (Renvela®) — Sevelamer Carbonate Tablets Dosed Three Times A Day

SUMMARY:
Approximately 45 hyperphosphatemic CKD patients not on dialysis will be entered into this study at approximately 20 sites within Europe and 5-10 in Australia. The purpose of this study is to determine if sevelamer carbonate tablets dosed three times a day (TID) is an effective treatment for the control of serum phosphorous levels in hyperphosphatemic CKD patients not on dialysis. Total length of participation is approximately 14 weeks.

ELIGIBILITY:
Inclusion Criteria:

* A minimum of 120 male and female patients with chronic kidney disease not requiring dialysis will be screened for participation in the study.
* Men or woman 18 years of age or older
* If currently taking phosphate binder(s), willing to stop this and enter a 2 week washout period
* Willing to avoid any intentional changes in diet such as fasting or dieting
* Have the following central laboratory measurements: 1. If not on a phosphate binder, a serum phosphorus measurement ≥ 5.5 mg/dL (1.76 mmol/L) at Screening (Visit1). 2. If taking a phosphate binder(s) at screening, a serum phosphorus measurement ≥ 5.5 mg/dL (1.76 mmol/L) after the two-week washout period at Visit 1a (Day 0).
* At Screening (Visit 1), have the following central laboratory measurements: 1. 25-hydroxyvitamin D ≥ 10 ng/mL 2. iPTH ≤ 800 pg/mL
* Willing and able to take sevelamer carbonate alone as a phosphate binder for the duration of the study
* Willing and able to maintain screening doses of lipid medication, 1,25 dihydroxyvitamin D, and/or cinacalcet for the duration of the study, except for safety reasons
* Willing and able to avoid antacids and phosphate binders containing aluminum, magnesium, calcium or lanthanum for the duration of the study unless prescribed as an evening calcium supplement
* If female and of childbearing potential (pre-menopausal and not surgically sterile), willing to use an effective contraceptive method throughout study, which includes barrier methods, hormones, or IUDs
* Expecting not to initiate dialysis for the duration of this study
* Considered compliant with phosphate binders (if applicable)
* Willing and able to provide informed consent
* Has not participated in any other investigational drug studies within 30 days prior to enrollment,
* Level of understanding and willingness to cooperate with all visits and procedures as described by the study personnel

Exclusion Criteria:

* Active bowel obstruction, dysphagia, swallowing disorder or severe gastrointestinal (GI) motility disorders
* Active ethanol or drug abuse, excluding tobacco use
* Use of anti-arrhythmic or anti-seizure medications for arrhythmia or seizure disorders.
* In the opinion of the investigator, patient has poorly controlled diabetes mellitus, poorly controlled hypertension, active vasculitis, HIV infection, or any clinically significant unstable medical condition
* Pregnant or breast-feeding
* Evidence of active malignancy except for basal cell carcinoma of the skin
* Unable to comply with the requirements of the study
* Known hypersensitivity to sevelamer or any constituents of the study drug
* Any other condition, which in the opinion of the investigator will prohibit the patient's inclusion in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2006-01; Primary Completion 2007-01 (Actual); Study Completion 2007-03 (Actual)

PRIMARY OUTCOMES:
Evaluate the efficacy of sevelamer carbonate tablets dosed three times per day (TID) with meals on control of serum phosphorus levels | Up to day 70
Evaluate the safety and tolerability of sevelamer carbonate tablets dosed TID with meals. | Up to day 70

SECONDARY OUTCOMES:
Serum calcium-phosphorus product | Up to day 70
Serum lipid profile [total cholesterol, high density lipoprotein (HDL) cholesterol, low density lipoprotein (LDL) cholesterol] | Up to day 70
Percent responders [serum phosphorus between 2.7 and 4.6 mg/dL (0.87 and 1.49 mmol/L) inclusive] at Day 56/ET | Up to day 70

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Genzyme, a Sanofi Company
Locations (25):
- Australia (5):
  - Nephrology Department, Princess Alexandra Hospital, Wooloongabba, Queensland
  - Renal Unit, The Queen Elizabeth Hospital, Woodville, South Australia
  - Renal Research Unit, Launceston General Hospital, Launceston, Tasmania
  - The Royal Melbourne Hospital, Department of Nephrology, Parkville, Victoria
  - Melbourne Renal Research Group, Epworth Medical Centre, Richmond, Victoria
- Denmark (4):
  - Nyremedicinsk Afdeling, Medicinerhuset, Aalborg
  - Medicinsk Afdeling, Copenhagen
  - Nefrologisk Afdeling, Hilleroed Sygehus, Hilleroed
  - Medicinsk Afdeling, nefrologisk, Roskilde Sygehus, Roskilde
- George Pompidou, European Hospital, Paris, France
- Germany (6):
  - Universitätsklinikum Aachen, Medizinsche Klinik II, Aachen
  - Universitätsklinikum Hamburg Eppendorf, Hamburg
  - Heimdialysezentrum, Heidelberg
  - KfH Nierenzentrum, Nuremberg
  - Stadt Klinken Solingen, Klinik für Nephrologie und Allgemeine Innere Medizin, Solingen
  - Nephrologisches Zentrum, Villingen-Schwenningen
- United Kingdom (9):
  - Birmingham Hospital, Queen Elizabeth Medical Centre, Birmingham, England
  - Southmead Hospital, Bristol, England
  - Addenbrooke's Dialysis Centre, Cambridge, England
  - Leicester General Hospital, Leicester, England
  - Renal Department, The Royal London Hospital, London, England
  - Renal & Urology SDU Offices, London, England
  - Renal Dialysis Unit, Manchester Royal Infirmary, Manchester, England
  - Department of Renal Medicine, Hope Hospital, Manchester, England
  - Renal Unit, Queen Alexandra Hospital, Portsmouth, England